CLINICAL TRIAL: NCT00181961
Title: A Dose-Finding Study of the Tolerability and Efficacy of Maca Root in Patients With Antidepressant-Induced Sexual Dysfunction
Brief Title: Safety and Effectiveness Study of Maca Root to Treat Antidepressant-Induced Sexual Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christina M. Dording, MD, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-P-001269
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Depression; Sexual Dysfunction
Keywords: antidepressant-induced sexual dysfunction
MeSH Terms: conditions — Depression; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Maca Root 1500mg (Experimental): Patients receiving 1500mg of maca root
  Interventions: Drug: Maca Root
- Maca Root 3000mg (Experimental): Patients receiving 3000mg of maca root
  Interventions: Drug: Maca Root

INTERVENTIONS:
Drug: Maca Root

SUMMARY:
The purpose of this study is to determine the dose of Maca Root effective for the treatment of antidepressant-induced sexual dysfunction in patients with DSM-IV defined Major Depressive Disorder. We propose to carry out a dose-finding pilot study to determine the minimum effective dose of Maca Root. We hypothesize that patients who receive Maca Root will experience alleviation of their sexual dysfunction, and this effect will be more pronounced in those who receive higher doses of maca root.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether Maca Root is effective for the treatment of antidepressant-induced sexual dysfunction, and to further determine whether higher doses of Maca Root powder would be more effective than lower doses in reducing the symptoms of antidepressant-induced sexual dysfunction. An additional aim of the study is to document the safety and tolerability of Maca Root, which could be particularly helpful in treating antidepressant-induced sexual dysfunction in elderly and cardiac-impaired populations taking oral nitrates who may not be eligible for treatment with the current oral phosphodiesterase inhibitors.

Subjects will be randomized into two arms of 10 for this 12-week study. The study will be double blind with regard to doses received. Ten subjects will receive 1500mg/day of maca for the 12-week period and the other 10 subjects will receive 3000mg/day of maca per day for the 12-week study period. Patients will be seen every other week. There is no placebo arm.

At the final study visit, week 12, subjects will be evaluated to see if their sexual function has returned.

After careful review of the literature we have found that there are very few studies that have evaluated Maca Root in humans. However the one very relevant study completed by Gonzalez and colleagues looked at doses of 1500 and 3000mg in men and found there were increased sexual interests on both doses. Thus, since this is a dose-finding study we believe this dose is an appropriate place to begin.

Hypotheses A:

The response rate will be higher for the high-dose maca group compared to the low-dose group; and this response will be comparable to the 50-85% reported with sildenafil.

Hypothesis B:

There will be a statistically significant difference in the magnitude of response between the two testing conditions, as measured by a decrease in baseline sexual dysfunction scores. The reduction in sexual dysfunction scores will be greater in the high-dose maca group than in the low-dose maca group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have been taking an SSRI, venlafaxine, nefazodone, or tri/hetero cyclic antidepressant for treatment of depression for at least 8 weeks, are currently at a stable dose of the antidepressant for at least 4 weeks, and have been consistently experiencing arousal dysfunction (inability to attain or maintain an adequate lubrication/swelling response of sexual excitement until completion of sexual activity) or orgasmic dysfunction (delayed orgasm/anorgasmia following a normal sexual excitement phase) that interferes with sexual function for at least 4 weeks.

Subjects must currently be euthymic (HAM-D< 10) and without significant anxiety symptoms (HAM-A<10). These scales will rely on retrospective reporting from the participant.

Subjects must have had no sexual dysfunction prior to taking an antidepressant and there must be a clear temporal relationship between the sexual dysfunction and the antidepressant treatment. Sexual dysfunction occurring as a symptom of the depressive disorder for which the antidepressant treatment was initiated is not considered to be a pre-existing condition under this definition.

* Subjects must meet at least one of the following criteria:

  * Inability to have an orgasm (anorgasmia), according to patient opinion
  * Clinically significant orgasm delay with masturbation or intercourse that according to patient opinion represents a meaningful delay and interferes with subject's sexual function compared with the subject's usual time to achieve orgasm in response to sexual stimulation prior to antidepressant medication
  * Inability to attain or maintain until completion of sexual activity an adequate an erection or lubrication swelling response of sexual excitement that, according to patient opinion, interferes with subject's sexual function, compared to prior to antidepressant medication.
  * Decreased libido according to patient opinion (and verified by objective measurements)
* Subjects must experience at least one of the above criterion items with distress and or disability.
* Subjects must be having or had been having some form of regular sexual activity (masturbation, oral sex, intercourse) at least twice monthly prior to the antidepressant treatment and are willing to continue efforts at sexual activity at least once weekly for the duration of the study
* Subjects must be in good general physical health

Exclusion Criteria:

* Primary or prior diagnosis of a sexual disorder (other than the side effect of the antidepressant drug or symptom of major depression)
* Sexual dysfunction secondary to general underlying medical condition
* Any uncontrolled psychiatric disorder
* Alcohol or substance abuse or dependence within the past six months
* Recent major relationship changes, disruption, or turmoil ongoing or anticipated which are unrelated to their sexual dysfunction
* Hamilton Depression and/or Anxiety Scale score (either) >10
* Blood pressure outside the range of 90/50 - 170/100
* Use of investigational drugs within prior 3 months or during study.
* Current use of other drugs for antidepressant induced sexual dysfunction or other therapies or medications to treat sexual dysfunction
* Hormone replacement therapy, unless patient has been on stable dose of hormone therapy for at least 3 months prior to the antidepressant treatment and had no sexual dysfunction while on the same hormone therapy regimen, and there is no change in the hormone replacement therapy during the study
* Pregnancy, lactating, or planning to become pregnant during the study
* Child bearing potential subjects unwilling and/or not prepared and/or who are judged unreliable to use an acceptable and verifiable form of contraception during the study
* Any clinically significant abnormality of the screening physical examination
* History of elevated PSA levels that are greater than 0.2 (as defined by MGH labs)
* History of prostate or other hormonal cancers
* Prior use of maca for at least two weeks
* Infection of the urogenital tract that may make sexual activity painful or difficult
* Subjects whose sexual partners are suffering from and/or receiving treatment for sexual dysfunction
* Receiving psychosexual or other therapy for sexual dysfunction and not willing to discontinue that treatment at screening
* Subjects not attempting some form of regular sexual activity at least twice monthly and at least once weekly during study visit intervals for the duration of the entire study
* Changes in antidepressant agent and/or dose of prescribed antidepressant agent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Dording, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Maca Root 1500mg: Patients receiving 1500mg of maca root
  Maca Root
- Maca Root 3000mg: Patients receiving 3000mg of maca root
  Maca Root
Period: Overall Study
Arm/Group | Maca Root 1500mg | Maca Root 3000mg
Started (Protocol defined enrolled as screened participants. Baseline visit determined randomization.) | 7 | 9
Completed | 6 | 4
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maca Root 1500mg | Maca Root 3000mg | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (12) | 34 (15) | 36 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 9 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Massachusetts General Hospital Sexual Dysfunction Inventory Scores
Description: Full title: Massachusetts General Hospital Sexual Dysfunction Inventory Minimum score for Men: 5 Minimum score for Women: 4 Maximum score for Men: 30 Maximum score for Women: 24
  *One item on the measure is for men only
  A score of a 5 (4 for women) indicates improvement in sexual function. A score of 10 (8 for women) indicates no change. A score higher than 10 (8 for women) indicates a level of sexual dysfunction.
Time Frame: baseline to endpoint (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Maca Root 1500mg | Maca Root 3000mg
Number analyzed (Participants) | 7 | 9
score on a scale | .249 (2.39) | .017 (1.15)
Statistical Analysis 1: Comparison: Maca Root 1500mg vs Maca Root 3000mg; Test type: Superiority; p = .016, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Maca Root 1500mg | Maca Root 3000mg
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 5/7 | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maca Root 1500mg (N=7) | Maca Root 3000mg (N=9)
GI Upset (Gastrointestinal disorders) | 2 (6) | 3 (4)
Headache (General disorders) | 0 (0) | 2 (2)
Irritability (General disorders) | 1 (1) | 1 (1)
Urinary Frequency (General disorders) | 0 (0) | 1 (2)
Sleep issues (General disorders) | 1 (3) | 0 (0)
Thicker Menstrual Discharge (General disorders) | 0 (0) | 1 (1)
Fibromyalgia Exacerbation (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No